CLINICAL TRIAL: NCT04642625
Title: Comparison of Ultrasound-guided Bilateral Erector Spinae Plane Block and Wound Infiltration for Spinal Surgical Analgesia
Brief Title: Comparison of Ultrasound-guided Bilateral ESP Block and Wound Infiltration for Spinal Surgical Analgesia
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Onur Kucuk, Department of anesthesiology and reanimation, Research Assistant, Trakya University
Other Study IDs: TÜTF-BAEK 2020/183
Record Dates: First submitted 2020-11-19; First posted 2020-11-24 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Pain, Postoperative; Spinal Disease; Anesthesia, Local; Anesthesia, Regional
Keywords: ultrasound-guided bilateral erector spina plane block; wound infiltration analgesia; spinal surgery
MeSH Terms: conditions — Pain, Postoperative; Spinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- wound infiltration analgesia: 25 patients who underwent wound infiltration analgesia
  Interventions: Other: Visual Analog Score; Other: patient satisfaction
- ultrasound-guided bilateral erector spina plan block analgesia: 25 patients who underwent ultrasound-guided bilateral erector spina plan block analgesia
  Interventions: Other: Visual Analog Score; Other: patient satisfaction
- wound infiltration and ultrasound-guided bilateral erector spina plan block analgesia both together: 25 patients who underwent wound infiltration and ultrasound-guided bilateral erector spina plan block analgesia
  Interventions: Other: Visual Analog Score; Other: patient satisfaction

INTERVENTIONS:
Other: Visual Analog Score — The VAS is a widely used tool in research and clinical practice, and its reliability and validity in pain assessment has been clearly demonstrated. It consists of a 100 mm line. 0 cm no pain, 10 cm is associated with 'worst possible pain'. The patient is asked to mark the line to 'score' the pain. VAS values of 1cm - 3cm weak, 4cm - 6cm moderate, and >7cm are the indicators of "severe pain".
  Other Names: VAS
Other: patient satisfaction — The patient's satisfaction with postoperative pain treatment will be recorded. 4 options; excellent, good, medium and bad.

SUMMARY:
The aim of our study is to determine the superior procedure in analgesia management by comparing the traditional wound infiltration technique with the ultrasound-guided bilateral erector spina plan block technique in spinal surgery patients.

DETAILED DESCRIPTION:
Patients in ASA I-II-III risk group aged 18-80 who will undergo spinal surgery by Trakya University Faculty of Medicine, Brain and Nerve Surgery will be included. In this study, patient data will be collected in the form of file scanning. Intra-operative; hemodynamic data of patients; heart rate, blood pressure values, anesthetic and other drugs applied, surgery and anesthesia durations will be written from the anesthesia document after the operation is over. In the study, the application preferred by the anesthesiologist for the patient will not be intervened. The patients will be divided into three groups; wound infiltration technique was applied, ultrasound-guided bilateral erector spina plan block technique was applied and both techniques were applied together. After the operation; pain values will be calculated by VAS at the 1st, 2nd, 4th, 6th, 12th and 24th hours of the patients. The patient's length of stay, satisfaction (excellent, good, moderate, poor) and methods used for analgesia will be recorded. With the results collected in our study, it will be determined which procedure is superior in pain management for spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective spine surgery
* No contraindication to the technique to be applied
* Not pregnant
* Being over the age of 18

Exclusion Criteria:

* Undergoing emergency spine surgery
* There is an obstacle to the technical process to be applied
* Pregnant patients
* Patients younger than 18 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in ASA I-II-III risk group aged 18-80 who will undergo spinal surgery by Trakya University Faculty of Medicine, Brain and Nerve Surgery will be included. 75 patients meeting these conditions will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Score | postoperative 24 hours score change
  It consists of a 100mm line. 0cm no pain, 10cm is associated with 'worst possible pain'. The patient is asked to mark a line to 'score' the pain. VAS values of 1cm-3cm weak, 4cm-6cm moderate, and >7cm are the indicators of "severe pain".After the operation; pain values will be calculated by VAS at the 1st, 2nd, 4th, 6th, 12th and 24th hours of the patients.

SECONDARY OUTCOMES:
patient satisfaction | postoperative 24 hours score change
  The patient's satisfaction with postoperative pain treatment will be recorded. 4 options; excellent, good, medium and bad.

CONTACTS AND LOCATIONS:
Overall Officials: SEVTAP HEKİMOĞLU ŞAHİN, Professor, Principal Investigator — Trakya University; ONUR KÜÇÜK, Resident, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Centrum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No